CLINICAL TRIAL: NCT01972451
Title: A Feasibility Randomised Controlled Trial (RCT) of Contrast Enhanced vs Non-enhanced Colonscopy in Index Bowel Cancer Screening to Reduce Bowel Cancer Mortality
Brief Title: Feasibility of Reduction in Right Sided Bowel Cancer Through Contrast Enhanced Colonoscopy
Acronym: CONSCOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lisette Nixon (Other)
Responsible Party: Sponsor-Investigator, Lisette Nixon, Senior Trial Manager, Cardiff University
Organization: Cardiff University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: WCTU065
Record Dates: First submitted 2013-10-07; First posted 2013-10-30 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colonoscopy without enhanced dye (Placebo Comparator): no enhanced dye
  Interventions: Procedure: Colonoscopy with enhanced dye
- Colonoscopy with enhanced dye (Active Comparator): enhanced dye
  Interventions: Procedure: Colonoscopy with enhanced dye

INTERVENTIONS:
Procedure: Colonoscopy with enhanced dye

SUMMARY:
The Bowel Cancer Screening program was implemented to address the important issue of prevention and early detection of bowel cancer. Results from the first few years of screening and previous smaller studies show that while in its current form it will save many lives, there continue to be polyps and cancers in the upper large bowel (right side) that may be difficult to detect. There is some evidence that these types of polyps (serrated polyps) may be at least partly responsible for cancers missed at the initial colonoscopy and have a faster rate of growth to cancer compared to conventional polyps (adenomas). We propose to examine participants undergoing screening colonoscopy with the addition of a contrast dye ( a safe food colouring agent base already used in various bowel camera procedures in standard clinical practice). This has been shown to improve detection of conventional polyps significantly even though it is considered by some to be more time consuming (possibly taking a few minutes longer) and requiring specific training to undertake. We hope to study the feasibility of undertaking these procedures to improve detection and removal of these polyps within the bowel screening program and potentially inform further studies to assess the impact of improved detection and consequent potentially reduced incidence of interval or missed bowel cancers in longer term follow up. Thus the main aims of this feasibility study are to assess if this type of procedure would be feasible to implement and acceptable to participants, colonoscopists and the screening program and also assess any additional time or costs involved to inform the question of if a larger study should then be undertaken to conclusively prove or disprove the merits of this approach in terms of health economics, cancer detection and survival.

ELIGIBILITY:
Inclusion Criteria:

* All participants testing positive on Faecal Occult Blood Test (FOBT) in the screening program who are eligible and appropriate for an index screening colonoscopy will be offered participation in the study.
* All participants attending for a one year surveillance colonoscopy if they have undergone an index screening colonoscopy as part of the study as per current guidelines for surveillance will also be offered inclusion

Exclusion Criteria:

* Any participants not deemed fit for colonoscopy on the screening program or undergoing alternative investigation such as CT Pneumocolon or minimal prep CT scan as their index procedure instead.
* Participants who have undergone previous colorectal surgery will be excluded from the study though their standard management in the screening program will continue unchanged.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1320 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Procedure time and withdrawal time | 1 year

SECONDARY OUTCOMES:
Number of people attending the screening | 1 year

OTHER OUTCOMES:
Colonoscopy procedure completeness | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Wales Cancer Trials Unit, Cardiff, United Kingdom

REFERENCES:
- [Derived] Hurt C, Ramaraj R, Farr A, Morgan M, Williams N, Philips CJ, Williams GT, Gardner G, Porter C, Sampson J, Hillier S, Heard H, Dolwani S; CONSCOP Clinical Research Consortium. Feasibility and economic assessment of chromocolonoscopy for detection of proximal serrated neoplasia within a population-based colorectal cancer screening programme (CONSCOP): an open-label, randomised controlled non-inferiority trial. Lancet Gastroenterol Hepatol. 2019 May;4(5):364-375. doi: 10.1016/S2468-1253(19)30035-4. Epub 2019 Mar 16. PMID 30885505
- See also: Sponsor study website — https://www.cardiff.ac.uk/centre-for-trials-research/research/studies-and-trials/view/conscop